CLINICAL TRIAL: NCT03456128
Title: Reducing Disability Following Hospital Discharge in Vulnerable Older Adults: The CAPABLE Intervention
Acronym: CAPABLE-VNSNY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00141968; 1R01AG056607-01 (NIH)
Record Dates: First submitted 2018-01-03; First posted 2018-03-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Disability Physical
Keywords: Older Adult; Rehospitalization; Physical function
MeSH Terms: interventions — CAPABLE protocol

STUDY DESIGN:
Intervention Model Description: The study is a single-masked, two-group, randomized trial to test the effectiveness of CAPABLE in reducing ADL difficulties compared to those randomized to usual care.
Who Masked: Outcomes Assessor
Masking Description: 1: 1. The outcome assessor will be unaware of which groups the older adults are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group will receive CAPABLE services. These include ≤10 sessions: ≤ 6 with an Occupational Therapist (OT) and ≤ 4 sessions with a Registered Nurse (RN) and up to ≤ $1,500 of home safety and home modifications from a licensed handyman who is guided by the OT. The OT and RN sessions will target participants' self-identified functional goals (e.g., getting safely into the tub, getting upstairs to sleep in own bed).
  Interventions: Other: CAPABLE
- Usual Care (No Intervention): Participants in the usual care group will not receive visit from study clinicians and will continue to receive their usual VNSNY CHOICE benefits and healthcare.

INTERVENTIONS:
Other: CAPABLE — It involves up to 10 in-home tailored interventions of approximately 60 minutes duration each over a 5-month period. The assessment driven interventions are delivered by an Occupational Therapist (OT) (≤ 6 home visits for ≤ 1hour), a Registered Nurse (RN) (≤ 4 home visits for ≤ 1hour), and a handyman (HM) team.
  Arms: Intervention

SUMMARY:
This study evaluates whether the utilization of integrated health services such as help with medications, muscle strengthening, balance training, pain management and home modification interventions can help improve older adults' ability to sleep, balance, walk, and take care of themselves after hospitalization.

DETAILED DESCRIPTION:
Currently, there is no evidence-based approach to improve post-hospitalization functional decline. CAPABLE uses a novel inter-professional team involving an occupational therapist, nurse, and handyman to improve ADLs in older adults post-hospitalization.

In a Center for Medicare & Medicaid Innovation (CMMI) demonstration project, CAPABLE demonstrated a 45% reduction of ADL difficulties in older adults from baseline to five months.The significance of this improvement could make the difference between aging at home independently and relocating to institutional care. While these results are encouraging, CAPABLE needs evaluation in real world health delivery contexts with more ethnic diversity.The purpose of this study is to test the effectiveness of CAPABLE in older adults in an active community health care program.

Interventions: CAPABLE Intervention: Participants in the treatment group will receive up to 10 in-home sessions (≤6 visits with an occupational therapist and ≤4 visits from a nurse)-and up to $1500 in safety and modification services from a licensed handyman. Each treatment participant will receive each intervention component (education, assessment, and identification of functional goals, specific strategies tailored to goals and based on protocols). Usual Care Group: Participants in the usual care group will not receive visit from study clinicians and will continue to receive their usual VNSNY CHOICE benefits and healthcare. After baseline, all study participants will be reassessed at 20 weeks and possibly a third interview at 52 weeks. Assessments will be completed by a research assistant masked to treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years old;
* Are 60 days post-hospitalization in an acute care setting and have had a Visiting Nurse Service of New York (VNSNY) visit;
* Have difficulty with at least one activity of daily living (ADL);
* Are a member of the VNSNY CHOICE Medicare Advantage Health Plan;
* Are able to stand with or without assistance; and
* Are available during the intervention period

Exclusion Criteria:

* Have significant cognitive impairment identified by the Callahan screening tool;
* Do not speak English or Spanish;
* Have had more than 3 hospitalizations within the past 12 months;
* Are actively receiving radiation or chemotherapy;
* Have plans to relocate in less than one year;
* Have diagnoses of the following: Dementia, Alzheimer's, Other Cerebral Degeneration, and serious cognitive impairment or OASIS assessment level 3 response on M1034 "serious progressive conditions that could lead to death within a year"

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 268 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Mean ADL Difficulty Score | 20-week follow-up period
  Change in ADL- the range is 0 - 16, with higher scores indicating that the participant needs a lot of help with performing many ADLs (is more disabled) and lower scores indicating that the participant is not disabled

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Szanton, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Visiting Nurse Service of New York, New York, New York, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03456128/Prot_SAP_003.pdf